CLINICAL TRIAL: NCT04845997
Title: NATIONAL VACCINATION REGISTRY FOR SARS-CoV-2 IN PATIENTS WITH RHEUMATIC DISEASES OF THE ARGENTINE SOCIETY OF RHEUMATOLOGY
Brief Title: COVID-19 Vaccination in Patients With Rheumatic Diseases
Acronym: SAR-CoVAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sociedad Argentina de Reumatologia (Other)
Responsible Party: Sponsor
Other Study IDs: 02
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Rheumatic Diseases
Keywords: SARS-CoV-2; COVID-19 Vaccines
MeSH Terms: conditions — Rheumatic Diseases | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: COVID-19 Vaccine — Patients with rheumatic diseases who have been vaccinated for COVID-19

SUMMARY:
The Argentine Society of Rheumatology (SAR) set out to develop a national register of patients with rheumatic diseases who have received a SARS-CoV-2 vaccine in order to assess their efficacy and safety in this population.

DETAILED DESCRIPTION:
This is an observational, longitudinal, multicenter study, including patients with rheumatic diseases who have been vaccinated for COVID-19 in Argentine or any country. Patients will be followed for 12 months and two evaluations will be performed, one at baseline and the other after the follow-up time is completed.

The aim of this registry is to evaluate the efficacy and safety of the SARS-CoV-2 vaccines in patients with rheumatic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age.
* Diagnosis of rheumatic disease treated or not with immunosuppressive agents
* Patients who have received at least one dose of a SARS-CoV-2 vaccine
* Signature of informed consent.

Exclusion Criteria:

* Patients who express their desire not to participate in the study or who are unable to give their informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatic diseases who have been vaccinated for COVID-19 in Argentine or any country
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
COVID-19 Vaccine efficacy | 12 month
  Number of patients who develop SARS-CoV-2 infection after vaccination
COVID-19 Vaccine safety | 12 month
  Number of patients who develop adverse events asssociated with vaccination

SECONDARY OUTCOMES:
New immunomediated events | 12 month
  Number of patients who develop new immunomediated events asssociated with vaccination. Description of the events.
Flare | 12 months
  Number of patients who develop a flare asssociated with vaccination. Description
Changes in the rheumatic disease treatment | 12 months
  Changes in the rheumatic disease treatment associated with vaccination, and study its influence on the efficacy (number of patients who develop SARS-CoV-2 infection after vaccination) and safety (number of patients who develop adverse events asssociated with vaccination) of the vaccine for SARS-CoV-2.
Vaccine efficacy among patients with immune mediated and non-immune mediated rheumatic diseases | 12 months
  Differences in the efficacy/safety profile of SARS-CoV-2 vaccine among patients with immune mediated and non-immune mediated rheumatic diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Isnardi, MD, Principal Investigator — Unidad de Investigación Sociedad Argentina Reumatología
Locations (2):
- Argentina (2):
  - Sociedad Argentina de Reumatología, Buenos Aires, Buenos Aires F.D.
  - Sociedad Argentina de Reumatologia, Buenos Aires

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Isnardi CA, Schneeberger EE, Kreimer JL, Luna PC, Echeverria C, Roberts K, de la Vega MC, Virasoro BM, Landi M, Quintana R, Exeni MED, Kogan N, Petkovic I, Pereira D, De Los Angeles Correa M, Zelaya MD, Tissera Y, Elkin MSG, Pisoni CN, Alonso C, Cogo AK, Cosatti MA, Garcia L, Retamozo C, de Los Angeles Severina M, Nieto RE, Rosemffet M, Mussano E, Bertoli A, Savio VG, Cosentino V, Pons-Estel GJ. An Argentinean cohort of patients with rheumatic and immune-mediated diseases vaccinated for SARS-CoV-2: the SAR-CoVAC Registry-protocol and preliminary data. Clin Rheumatol. 2022 Oct;41(10):3199-3209. doi: 10.1007/s10067-022-06253-5. Epub 2022 Jun 28. PMID 35760939